CLINICAL TRIAL: NCT03303989
Title: REduCing Immunogenicity to PegloticasE (RECIPE) Study
Acronym: RECIPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 300000591
Record Dates: First submitted 2017-09-29; First posted 2017-10-06 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Gout Chronic
MeSH Terms: interventions — Pegloticase

STUDY DESIGN:
Intervention Model Description: Phase II, double blind, placebo controlled multisite proof-of-concept trial in subjects initiating pegloticase for treatment of chronic gout
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pegloticase + MMF (Experimental): Participants randomized to this arm will receive pegloticase + mycophenolate mofetil.
  Interventions: Drug: Pegloticase 8 MG/ML [Krystexxa]; Drug: MMF
- pegloticase + placebo (Placebo Comparator): Participants randomized to this arm will receive pegloticase + placebo
  Interventions: Drug: Placebo; Drug: Pegloticase 8 MG/ML [Krystexxa]

INTERVENTIONS:
Drug: Pegloticase 8 MG/ML [Krystexxa] — Participants randomized to the pegloticase + MMF arm will start two week run-in on 1) mycophenolate mofetil at 500 mg/BID or the first week, titrating dose up to 1000mg/BID for the second week of run-in prior to the first infusion; and 2) Pegloticase 8 mg IV every two weeks following 2 week run-in period, Mycophenolate mofetil therapy will continue for 12 weeks at the highest tolerated dose. After the 12-week combination mycophenolate mofetil and pegloticase study period, participants will continue open label pegloticase therapy for an additional three months.
  Other Names: Krystexxa
  Arms: pegloticase + MMF
Drug: MMF — Participants randomized to the pegloticase + MMF arm will start two week run-in on 1) mycophenolate mofetil at 500 mg/BID or the first week, titrating dose up to 1000mg/BID for the second week of run-in prior to the first infusion; and 2) Pegloticase 8 mg IV every two weeks following 2 week run-in period, Mycophenolate mofetil therapy will continue for 12 weeks at the highest tolerated dose. After the 12-week combination mycophenolate mofetil and pegloticase study period, participants will continue open label pegloticase therapy for an additional three months.
  Other Names: Cell Cept
  Arms: pegloticase + MMF
Drug: Placebo — Participants randomized to the pegloticase + placebo arm will start two week run-in on 1) placebo at 500 mg/BID or the first week, titrating dose up to 1000mg/BID for the second week of run-in prior to the first infusion; and 2) Pegloticase 8 mg IV every two weeks following 2 week run-in period. After the 12-week combination placebo and pegloticase study period, participants will continue open label pegloticase therapy for an additional three months.
  Arms: pegloticase + placebo
Drug: Pegloticase 8 MG/ML [Krystexxa] — Participants randomized to the pegloticase + placebo arm will start two week run-in on 1) placebo at 500 mg/BID or the first week, titrating dose up to 1000mg/BID for the second week of run-in prior to the first infusion; and 2) Pegloticase 8 mg IV every two weeks following 2 week run-in period. After the 12-week combination placebo and pegloticase study period, participants will continue open label pegloticase therapy for an additional three months.
  Other Names: Krystexxa
  Arms: pegloticase + placebo

SUMMARY:
Pegloticase treatment for chronic refractory gout is limited by immunogenicity. The investigators propose the REduCing Immunogenicity to PegloticasE (RECIPE) trial to begin to investigate the question of whether a short course of immune modulating therapy with mycophenolate mofetil can significantly and safely attenuate immunogenicity to pegloticase and ensure patients afflicted with chronic refractory gout have better treatment outcomes and improved quality of life.

DETAILED DESCRIPTION:
Pegloticase is highly efficacious therapy for chronic refractory gout patients (n = > 400K in the US alone). It decreases serum urate (sUA) levels to often undetectable levels and reduces tophi burden. However, its long-term real world effectiveness is severely limited due to its immunogenicity caused by anti-pegloticase antibody formation. REducing Immunogenicity to PEgloticase (RECIPE) is a Phase II, double-blind, placebo controlled, proof-of-concept trial in 32 subjects initiating pegloticase for treatment of chronic refractory gout. RECIPE will investigate the preliminary efficacy and safety of using immune modulating therapy with mycophenolate mofetil (MMF) to prevent immunogenicity conferred by pegloticase. Subjects will be randomized 3:1 to receive MMF vs. placebo in addition to everyone receiving pegloticase. The co-primary aims of the RECIPE trial are to 1) determine if a 12 week course of immune modulating therapy with daily MMF can safely and significantly attenuate immunogenicity to pegloticase as determined by the proportion of participants achieving and maintaining an sUA less than or equal to 6 mg/dL through 12 weeks, compared to concurrent controls, and 2) to assess the incidence and types of adverse events and infusion reaction. After 12 weeks of co-administration, all participants will continue on pegloticase for an additional 12 weeks without combination MMF immune modulating therapy to evaluate the longer term benefits (durability) and safety of this approach. The secondary aims are to: 1) Determine the 6 month durability of immune modulation after discontinuation of the short course of MMF by: a) assessing the absolute change in sUA from baseline to Week 24, and Week 12 to Week 24 and b) determining the proportion of participants with sUA ≤ 6 mg/dL through 24 weeks, and Week 12 to Week 24; 2) Identify and characterize the pegloticase immune response by immunoglobulin isotypes (IgG and IgM), specificities, and antibody titer; and 3) Examine patient reported outcomes (PROs) using the NIH supported Patient Reported Outcomes Measurement Information System (PROMIS) and Gout Impact Scale (GIS) instruments. The University of Alabama at Birmingham (UAB) and the University of Michigan (UM), two large academic gout and immunology research centers, which in aggregate see nearly 10,000 gout patients annually, will serve as the two lead study sites and are very well-positioned to address the clinical and immunologic questions posed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years of age
* Diagnosed with chronic refractory gout*

  * Defined as: Persons whose signs and symptoms are inadequately controlled with urate lowering therapy (e.g. xanthine oxidase inhibitors or uricosuric agents) at a medically appropriate dose or for whom these drugs are contraindicated.

Exclusion Criteria:

* Any serious acute bacterial infection (2 weeks prior to Visit 1), unless treated and completely resolved with antibiotics
* Severe chronic or recurrent bacterial infections (such as recurrent pneumonia, chronic bronchiectasis)
* Current immunocompromised condition, including current or chronic treatment with immunosuppressive agents
* Subjects at risk for tuberculosis. Specifically, subjects with: i) current clinical, radiographic or laboratory evidence of active or latent TB; ii) a history of active TB within the last 3 years even if it was treated; iii) a history of active TB greater than 3 years ago unless there is documentation that the prior anti-TB treatment was appropriate in duration and type
* Known Hepatitis B surface antigen-positive or Hepatitis B DNA positive subjects
* Known Hepatitis C RNA-positive subjects
* Human Immunodeficiency Virus (HIV) infection
* G6PD deficiency (tested at Screening Visit 1)
* Severe chronic renal impairment (glomerular filtration rate [GFR] <25 mL/min/1.73 m2) or currently on dialysis
* Subjects having any transplant surgery requiring maintenance immunosuppressive therapy
* Non-compensated congestive heart failure, uncontrolled arrhythmia, treatment for acute coronary syndrome (myocardial infarction or unstable angina), or hospitalization for congestive heart failure within 3 months of screening or uncontrolled blood pressure (>160/100 mm Hg) at baseline (Screening Visit 1 and Week 0/Baseline visits)
* Participants who are pregnant, planning to become pregnant, breastfeeding, or not on an effective form of birth control (defined in Study Protocol section 7.1)
* Prior treatment with pegloticase, another recombinant uricase, or concomitant therapy with a polyethylene glycol (PEG)-conjugated drug
* Known allergy to pegylated products or history of anaphylactic reaction to a recombinant protein or porcine product
* Subjects in whom MMF treatment is contraindicated or considered inappropriate
* Recipient of an investigational drug within 4 weeks prior to study drug administration or plans to take an investigational agent during the study
* Current liver disease as determined by alanine transaminase ALT or aspartate transaminase (AST) levels >3 times upper limit of normal
* Currently receiving treatment for ongoing cancer, excluding non-melanoma skin cancer
* History of malignancy within 5 years other than skin cancer or in situ carcinoma of cervix
* Uncontrolled hyperglycemia with a plasma glucose value >240 mg/dL at screening
* Diagnosed osteomyelitis
* Individuals with hypoxanthine-guanine phosphoribosyl-transferase (HGPRT) deficiency such as Lesch-Nyhan and Kelley-Seegmiller syndrome
* Not good candidate for the study based on opinion of the Investigator (e.g., cognitive impairment) that might create undue risk to the participant or interfere with the participant's ability to comply with the protocol requirements, or to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Saag, MD, Principal Investigator — Professor
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khanna PP, Khanna D, Cutter G, Foster J, Melnick J, Jaafar S, Biggers S, Rahman AKMF, Kuo HC, Feese M, Kivitz A, King C, Shergy W, Kent J, Peloso PM, Danila MI, Saag KG. Reducing Immunogenicity of Pegloticase With Concomitant Use of Mycophenolate Mofetil in Patients With Refractory Gout: A Phase II, Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Rheumatol. 2021 Aug;73(8):1523-1532. doi: 10.1002/art.41731. Epub 2021 May 19. PMID 33750034

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegloticase + MMF | Pegloticase + Placebo
Started | 24 | 11
Completed | 22 | 10
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: 35 participants were randomized. Three participants withdrew after randomization, but prior to first pegloticase infusion. Baseline characteristics are of the 32 participants (22 in MMF+Peg, 10 in PBO+Peg)
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegloticase + MMF | Pegloticase + Placebo | Total
Number analyzed (Participants) | 22 | 10 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (9.4) | 55.5 (10.7) | 55.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 19 | 9 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 10 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 0 | 5
  White | 15 | 10 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 10 | 32
American College of Rheumatology / European League Against Rheumatism Flare Criteria Score [Mean (Standard Deviation); unit: Score on a scale] — Maximum score is 23 points across 3 domains. Score of >=8 classifies a subject as having gout
  Domains include 1) clinical parameters, 2) laboratory parameters and 3) imaging parameters. The specific domains and their respective definitions are available at https://ard.bmj.com/content/74/10/1789. Domains were designed to be scored based on the totality of the subjects' symptomatic disease experience. Categories within domains are hierarchical and mutually exclusive, such that if a higher and a lower category have been fulfilled at different points in time, the higher one should be scored.
  Score on a scale | 13.5 (2.8) | 13.8 (2.7) | 13.5 (2.6)
Gout Flare History (flare within the last year) [Count of Participants; unit: Participants]
  Yes | 15 | 5 | 20
  No | 7 | 5 | 12
Duration of Gout [Mean (Standard Deviation); unit: years] | 13.3 (9.8) | 13.4 (7.4) | 13.4 (9.0)
PROMIS Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — The higher score the more severity PROMIS Pain scores raw ranges from 3 to 15 (convert to T-Score as minimum: 30.7 and maximum: 71.8)
  units on a scale | 50.8 (11.3) | 45.0 (12.4) | 49.0 (11.8)
PROMIS Physical Function [Mean (Standard Deviation); unit: units on a scale] — Higher score worse outcome. PROMIS Physical Function raw ranges from 4 to 20 (convert to minimum: 22.9 and maximum: 56.9)
  units on a scale | 37.5 (7.8) | 33.8 (6.4) | 36.3 (8.6)
Gout Impact Score [Mean (Standard Deviation); unit: Score on a scale] — The gout impact score is a disease-specific measure that adequately captures the impact of gout over time, and allows patients to describe the impact of gout on their health related quality of life.
  24 item questionnaire with responses on Likert-type scales (e.g., strongly agree to strongly disagree; all of the time to none of the time).The higher score the more severity. Score range: 0-96.
  Score on a scale | 45.7 (7.5) | 46.4 (7.1) | 45.9 (7.3)
Serum Urate Level [Mean (Standard Deviation); unit: mg/dL] | 8.9 (1.8) | 9.8 (1.3) | 9.2 (1.7)
Body Mass Index [Count of Participants; unit: Participants]
  25 to < 30 | 3 | 1 | 4
  30 to < 45 | 18 | 7 | 25
  ≥45 | 1 | 2 | 3
Comorbidities [Count of Participants; unit: Participants]
  Diabetes Mellitus /Metabolic Syndrome: Yes | 3 | 2 | 5
  Diabetes Mellitus /Metabolic Syndrome: No | 19 | 8 | 27
  Cerebral Vascular Vascular Disease/Heart Accident/Peripheral Vascular Disease: Yes | 8 | 6 | 14
  Cerebral Vascular Vascular Disease/Heart Accident/Peripheral Vascular Disease: No | 14 | 4 | 18
  Systemic Hypertension: Yes | 18 | 7 | 25
  Systemic Hypertension: No | 4 | 3 | 7
  Dyslipidemia: Yes | 8 | 4 | 12
  Dyslipidemia: No | 14 | 6 | 20
  Kidney Stones: Yes | 4 | 5 | 9
  Kidney Stones: No | 18 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving and Maintaining an sUA ≤ to 6 Milligram Per Deciliter (mg/dL) Through 12 Weeks
Description: Proportion of participants achieving and maintaining an sUA ≤ to 6 mg/dL through 12 weeks, compared to concurrent controls.
Time Frame: 12 weeks
Population: 32 participants received at least one dose of pegloticase and were included in modified intention-to-treat analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegloticase + MMF | Pegloticase + Placebo
Number analyzed (Participants) | 22 | 10
Participants
  Yes | 19 | 4
  No | 3 | 6
Statistical Analysis 1: Comparison: Pegloticase + MMF vs Pegloticase + Placebo; Fisher's exact tests were performed to compare baseline and clinical characteristics between treatment groups as appropriate; Test type: Superiority — Efficacy of MMF was examined by the proportion of responders in MMF+Peg compared to PBO+Peg. Rates of the primary outcome were compared using proportions and 95% confidence intervals and tested for differences using Fisher's exact test; p < 0.01, Fisher Exact

ADVERSE EVENTS:
Time Frame: 36 weeks
Description: Adverse event was defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related. Adverse Events were monitored/assessed based on organ system class.
Arm/Group | Pegloticase + MMF | Pegloticase + Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/22 | 1/10
Other Adverse Events (participants affected / at risk) | 15/22 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegloticase + MMF (N=22) | Pegloticase + Placebo (N=10)
Infusion Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Motor Vehicle Crash (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegloticase + MMF (N=22) | Pegloticase + Placebo (N=10)
Cardia (Cardiac disorders) | 2 (2) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 4 (4) | 1 (1)
Infections (Infections and infestations) | 2 (2) | 0 (0)
Musculoskeletal (arthralgia, myalgia, low back pain, orthopedic trauma, bursitis tendonitis) (Musculoskeletal and connective tissue disorders) | 9 (19) | 1 (2)
Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Other (Lab abnormality, anxiety, neurological, and oral pain) (General disorders) | 9 (11) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT03303989/Prot_SAP_ICF_000.pdf